CLINICAL TRIAL: NCT00279682
Title: Prevention of Suicide in Primary Care Elderly: Collaborative Trial
Brief Title: Prevention of Suicide in Primary Care Elderly: Collaborative Trial (PROSPECT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: University of Pennsylvania (Other); University of Pittsburgh (Other); National Institute of Mental Health (NIMH) (NIH); Forest Laboratories (Industry); The John A. Hartford Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH059366 (NIH); R01MH059380 (NIH); R01MH059381 (NIH)
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2006-01-19 (Estimated); Status verified 2006-01

CONDITIONS: Depression; Suicide, Attempted
Keywords: depression; suicide; geriatric; elderly; primary care
MeSH Terms: conditions — Depression; Suicide, Attempted; Suicide

INTERVENTIONS:
Behavioral: treatment guidelines and depression care management

SUMMARY:
The purpose of this study was to determine the effect of a primary care intervention on reducing suicidal ideation and depression in older patients.

DETAILED DESCRIPTION:
Suicide rates are highest in late life; the majority of older adults who die by suicide have seen a primary care physician in preceding months. Depression is the strongest risk factor for late-life suicide and for suicide's precursor, suicidal ideation.

The aim of the study was to determine the extent to which an intervention taht combined treatment guidelines with care management reduced rates of depression and suicide ideation in older primary care patients. The study randomized 20 primary care practices from New York City, Philadelphia, and Pittsburgh regions into intervention or usual car. The used a two-stage sampling design that resulted in a representative sample with an oversample of depressed patients (total n=1238 subjects including 598 with a depression diagnosis and 640 with no depression diagnosis). Patients were assessed at baseline, 4, 8, 12, 18 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

upcoming appointment with primary care clinician

Exclusion Criteria:

* inability to give consent
* minimental status examination <18
* ability to communicate in English

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200
Dates: Start 1999-05; Study Completion 2003-08

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale
Scale for Suicide Ideation

SECONDARY OUTCOMES:
All cause and cause-specific mortality
disability (Sf12; instrumental activities of daily living)

CONTACTS AND LOCATIONS:
Overall Officials: George S Alexopoulos, MD, Principal Investigator — Weill Medical College of Cornell University; Ira Katz, MD. Ph.D., Principal Investigator — University of Pennsylvania; Charles F Reynolds, MD, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - Weill Medical College of Cornell University, White Plains, New York
  - Universilty of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Bruce ML, Pearson JL. Designing an intervention to prevent suicide: PROSPECT (Prevention of Suicide in Primary Care Elderly: Collaborative Trial). Dialogues Clin Neurosci. 1999 Sep;1(2):100-12. doi: 10.31887/DCNS.1999.1.2/mbruce. PMID 22033641
- [Result] Bruce ML, Ten Have TR, Reynolds CF 3rd, Katz II, Schulberg HC, Mulsant BH, Brown GK, McAvay GJ, Pearson JL, Alexopoulos GS. Reducing suicidal ideation and depressive symptoms in depressed older primary care patients: a randomized controlled trial. JAMA. 2004 Mar 3;291(9):1081-91. doi: 10.1001/jama.291.9.1081. PMID 14996777
- [Result] Alexopoulos GS, Katz IR, Bruce ML, Heo M, Ten Have T, Raue P, Bogner HR, Schulberg HC, Mulsant BH, Reynolds CF 3rd; PROSPECT Group. Remission in depressed geriatric primary care patients: a report from the PROSPECT study. Am J Psychiatry. 2005 Apr;162(4):718-24. doi: 10.1176/appi.ajp.162.4.718. PMID 15800144
- [Result] Gallo JJ, Bogner HR, Morales KH, Post EP, Ten Have T, Bruce ML. Depression, cardiovascular disease, diabetes, and two-year mortality among older, primary-care patients. Am J Geriatr Psychiatry. 2005 Sep;13(9):748-55. doi: 10.1176/appi.ajgp.13.9.748. PMID 16166403
- [Derived] Gallo JJ, Hwang S, Truong C, Reynolds CF, Spira AP. Role of persistent and worsening sleep disturbance in depression remission and suicidal ideation among older primary care patients: the PROSPECT study. Sleep. 2020 Oct 13;43(10):zsaa063. doi: 10.1093/sleep/zsaa063. PMID 32239161
- [Derived] Gilman SE, Fitzmaurice GM, Bruce ML, Ten Have T, Glymour MM, Carliner H, Alexopoulos GS, Mulsant BH, Reynolds CF 3rd, Cohen A. Economic inequalities in the effectiveness of a primary care intervention for depression and suicidal ideation. Epidemiology. 2013 Jan;24(1):14-22. doi: 10.1097/EDE.0b013e3182762403. PMID 23232609
- [Derived] Bao Y, Alexopoulos GS, Casalino LP, Ten Have TR, Donohue JM, Post EP, Schackman BR, Bruce ML. Collaborative depression care management and disparities in depression treatment and outcomes. Arch Gen Psychiatry. 2011 Jun;68(6):627-36. doi: 10.1001/archgenpsychiatry.2011.55. PMID 21646579
- [Derived] Alexopoulos GS, Reynolds CF 3rd, Bruce ML, Katz IR, Raue PJ, Mulsant BH, Oslin DW, Ten Have T; PROSPECT Group. Reducing suicidal ideation and depression in older primary care patients: 24-month outcomes of the PROSPECT study. Am J Psychiatry. 2009 Aug;166(8):882-90. doi: 10.1176/appi.ajp.2009.08121779. Epub 2009 Jun 15. PMID 19528195